CLINICAL TRIAL: NCT03320330
Title: A Phase 1/2 Study of VX15/2503 in Children, Adolescents, or Young Adults With Recurrent or Relapsed Solid Tumors
Brief Title: Pepinemab in Treating Younger Patients With Recurrent, Relapsed, or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADVL1614; NCI-2017-01103 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ADVL1614 (Other: Pediatric Early Phase Clinical Trial Network); ADVL1614 (Other: CTEP); UM1CA097452 (NIH)
Record Dates: First submitted 2017-10-13; First posted 2017-10-25 (Actual); Results first posted 2022-04-26 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Recurrent Malignant Solid Neoplasm; Recurrent Osteosarcoma; Refractory Malignant Solid Neoplasm; Refractory Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — pepinemab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pepinemab) (Experimental): Patients receive pepinemab IV over 60 minutes on days 1 and 15. Treatment repeats every 28 days for 13 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pepinemab; Other: Pharmacological Study

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pepinemab — Given IV
  Other Names: moAb VX15/2503; VX15/2503
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects and best dose of pepinemab and to see how well it works in treating younger patients with solid tumors that have come back after treatment, or do not respond to treatment. Immunotherapy with monoclonal antibodies, such as pepinemab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) and/or recommended phase 2 dose of pepinemab (VX15/2503) administered as an intravenous infusion every 14 days to children with recurrent or refractory solid tumors. (Part A) II. To define and describe the toxicities of VX15/2503 administered on this schedule. (Parts A-B) III. To characterize the pharmacokinetics of VX15/2503 in children with recurrent or refractory cancer. (Parts A-B) IV. To preliminarily define the antitumor activity of VX15/2503 for the treatment of relapsed or refractory osteosarcoma. (Part B) V. To determine if VX15/2503 either improves the disease control rate at 4 months in patients with recurrent measurable osteosarcoma or produces an objective response rate in patients with relapsed or refractory osteosarcoma. (Part B)

SECONDARY OBJECTIVES:

I. To assess the pharmacodynamics of VX15/2503 through VX15/2503 saturation of T-lymphocytes.

II. To assess the immunogenicity of VX15/2503 in pediatric patients with recurrent or refractory cancer.

EXPLORATORY OBJECTIVES:

I. To evaluate potential biomarkers of VX15/2503 sensitivity including SEMA4D, PlexinB1, and other markers of immune cell infiltration in archival tumor tissues.

OUTLINE: This is a phase I, dose-escalation study followed by a phase II study.

Patients receive pepinemab intravenously (IV) over 60 minutes on days 1 and 15. Treatment repeats every 28 days for 13 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Part A: Patients with recurrent or refractory solid tumors are eligible, excluding central nervous system (CNS) tumors; patients must have had histologic verification of malignancy at original diagnosis or relapse
* Part B: Patients with recurrent or refractory osteosarcoma are eligible; patients must have had histologic verification of malignancy at original diagnosis or relapse
* Part A: Patients must have either measurable or evaluable disease
* Part B: Patients must have measurable disease
* Patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment; if after the required timeframe, the numerical eligibility criteria are met, e.g. blood count criteria, the patient is considered to have recovered adequately

  * Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive

    * >= 21 days after the last dose of cytotoxic or myelosuppressive chemotherapy (42 days if prior nitrosourea)
  * Anti-cancer agents not known to be myelosuppressive (e.g. not associated with reduced platelet or absolute neutrophil count [ANC] counts): >= 7 days after the last dose of agent
  * Antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1
  * Corticosteroids: If used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
  * Hematopoietic growth factors: >= 14 days after the last dose of a long-acting growth factor (e.g. pegfilgrastim) or 7 days for short-acting growth factor; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair and the study-assigned research coordinator
  * Interleukins, interferons and cytokines (other than hematopoietic growth factors): >= 21 days after the completion of interleukins, interferon or cytokines (other than hematopoietic growth factors)
  * Stem cell Infusions (with or without total body irradiation [TBI]):

    * Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including donor lymphocyte infusion (DLI) or boost infusion: >= 84 days after infusion and no evidence of graft versus host disease (GVHD)
    * Autologous stem cell infusion including boost infusion: >= 42 days
  * Cellular Therapy: >= 42 days after the completion of any type of cellular therapy (e.g. modified T cells, natural killer [NK] cells, dendritic cells, etc.)
  * Radiation Therapy (XRT)/External Beam Irradiation including Protons: >= 14 days after local XRT; >= 150 days after TBI, craniospinal XRT or if radiation to >= 50% of the pelvis; >= 42 days if other substantial bone marrow (BM) radiation
  * Radiopharmaceutical therapy (e.g., radiolabeled antibody, 131I-MIBG): >= 42 days after systemically administered radiopharmaceutical therapy
* Patients must not have received prior exposure to VX15/2503
* Peripheral absolute neutrophil count (ANC) >= 1000/mm^3
* Platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
* Hemoglobin >= 8.0 g/dL at baseline (may receive red blood cell [RBC] transfusions)
* Patients with known bone marrow metastatic disease will be eligible for study provided they meet the blood counts above (may receive transfusions provided they are not known to be refractory to red cell or platelet transfusions); these patients will not be evaluable for hematologic toxicity; at least 5 of every cohort of 6 patients must be evaluable for hematologic toxicity for the dose-escalation part of the study; if dose-limiting hematologic toxicity is observed, all subsequent patients enrolled must be evaluable for hematologic toxicity
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 ml/min/1.73 m^2 or
* A serum creatinine based on age/gender as follows:

  * Age: 1 to < 2 years; Male: 0.6 mg/dL; Female: 0.6 mg/dL
  * Age: 2 to < 6 years; Male: 0.8 mg/dL; Female: 0.8 mg/dL
  * Age: 6 to < 10 years; Male: 1 mg/dL; Female: 1 mg/dL
  * Age: 10 to < 13 years; Male: 1.2 mg/dL; Female: 1.2 mg/dL
  * Age: 13 to < 16 years; Male: 1.5 mg/dL; Female: 1.4 mg/dL
  * Age: >= 16 years; Male: 1.7 mg/dL; Female: 1.4 mg/dL
* Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age
* Alanine aminotransferase (ALT) serum glutamic pyruvic transaminase (SGPT) =< 135 U/L; for the purpose of this study, the ULN for ALT is 45 U/L
* Serum albumin >= 2 g/dL
* No clinical indications such as evidence of dyspnea at rest, or exercise intolerance due to pulmonary insufficiency
* If clinical indications, pulse oximetry > 94% on room air
* All patients and/or their parents or legally authorized representatives must sign a written informed consent; assent, when appropriate, will be obtained according to institutional guidelines
* Tissue blocks or slides must be sent; if tissue blocks or slides are unavailable, the study chair must be notified prior to enrollment

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study; pregnancy tests must be obtained in girls who are post-menarchal; males or females of reproductive potential may not participate unless they have agreed to use two effective methods of birth control, including a medically accepted barrier or contraceptive method (e.g., male or female condom) for the duration of the study; abstinence is an acceptable method of birth control
* Patients receiving systemic corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible; if used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of systemic corticosteroid; Note: patients who are using topical or inhaled corticosteroids are eligible
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anti-cancer agents are not eligible (except leukemia patients receiving hydroxyurea, which may be continued until 24 hours prior to start of protocol therapy)
* Patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial
* Patients who have an uncontrolled infection are not eligible
* Patients who have received a prior solid organ transplantation are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible

Ages: 12 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily G Greengard, Principal Investigator — COG Phase I Consortium
Locations (24):
- United States (24):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Derived] Greengard E, Williams R, Moriarity B, Liu X, Minard CG, Reid JM, Fisher T, Evans E, Pastore DR, Zauderer M, Voss S, Fox E, Weigel BJ. A phase 1/2 study of pepinemab in children, adolescents, or young adults with recurrent or refractory solid tumors: A children's oncology group consortium report (ADVL1614). Pediatr Blood Cancer. 2024 Jun;71(6):e30938. doi: 10.1002/pbc.30938. Epub 2024 Mar 23. PMID 38520670
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A Phase I/II Study of VX15/2503 in Children, Adolescents, or Young Adults with Recurrent or Relapsed Solid Tumors. This trial studies the side effects and best dose of pepinemab to see how well it works in treating younger patients that have come back after treatment, or do not respond to treatment. Immunotherapy with monoclonal antibodies, such as pepinemab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.
Pre-assignment Details: Part A (phase 1) portion of the study was to determine if Dose Level 1 (DL1), 20mg/kg pepinemab, was the Maximum Tolerated Dose (MTD)/Recommended Phase 2 Dose (RP2D). There were no dose levels above DL1. However, there was a possible lower dose level of 10mg/kg pepinemab if DL1 was too toxic. Since were no patients with dose-limiting toxicities, all patients in Part A PK (Expansion) and Part B (phase 2) received 20mg/kg pepinemab
Groups:
- Part A: 20 mg/kg (Phase 1); Part A PK: 20 mg/kg (Expansion): Patients ≥ 12 months and ≤ 21 years of age with recurrent or refractory solid tumors, excluding CNS tumors, receive 20 mg/kg of pepinemab IV over 60 minutes on days 1 and 15. Treatment repeats every 28 days for 13 cycles in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies Pepinemab: Given IV Pharmacological Study: Correlative studies
- Part B: 20 mg/kg (Phase 2): Patients ≥ 12 months and ≤ 30 years with recurrent or refractory osteosarcoma, receive 20 mg/kg of pepinemab IV over 60 minutes on days 1 and 15. Treatment repeats every 28 days for 13 cycles in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies Pepinemab: Given IV Pharmacological Study: Correlative studies
Period: Overall Study
Arm/Group | Part A: 20 mg/kg (Phase 1) | Part A PK: 20 mg/kg (Expansion) | Part B: 20 mg/kg (Phase 2)
Started | 6 | 6 | 14
Completed | 0 | 1 | 0
Not Completed | 6 | 5 | 14
Not completed — Lack of Efficacy | 5 | 5 | 14
Not completed — Physician Decision | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part A; Part A PK; Part B: Patients must be ≥ 12 months and ≤ 21 years of age, recurrent or refractory solid tumors are eligible, excluding CNS tumors.
- Total: Total of all reporting groups
Arm/Group | Part A | Part A PK | Part B | Total
Number analyzed (Participants) | 6 | 6 | 14 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 6 | 6 | 16
  Between 18 and 65 years | 2 | 0 | 8 | 10
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Year] | 17.5 (2.3) | 7.7 (4.2) | 17.4 (7.1) | 15.2 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 8 | 12
  Male | 4 | 4 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 4 | 6
  Not Hispanic or Latino | 5 | 4 | 8 | 17
  Unknown or Not Reported | 0 | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 3
  White | 2 | 3 | 7 | 12
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 1 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities
Description: Frequency (%) of patients with dose limiting toxicities by dose level and study part.
Time Frame: Up to 28 days
Population: The patients who had DLT in dose escalation course.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: 20 mg/kg (Phase 1) | Part A PK: 20 mg/kg (Expansion) | Part B: 20 mg/kg (Phase 2)
Number analyzed (Participants) | 6 | 6 | 14
Participants | 0 | 0 | 1
Statistical Analysis 1: Comparison: Part A: 20 mg/kg (Phase 1); Test type: Other — Recommended Phase 2 dose of pepinemab (VX15/2503), administered to children with recurrent or refractory solid tumors (Part A), was determined by the rolling-6 design; Recommended Phase 2 dose = 20 — Recommended Phase 2 dose of pepinemab (VX15/2503) is 20 mg/kg

2. Primary Outcome: Patients Who Had Grade 3 or Above Toxicities With the Three Attributions, 'DEFINITE', 'POSSIBLE','PROBABLE'
Description: Frequency of patients experiencing at least grade 3 toxicity according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 by dose level and study part.
Time Frame: Up to 28 days
Population: Part A and B Patients
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: 20 mg/kg (Phase 1) | Part A PK: 20 mg/kg (Expansion) | Part B: 20 mg/kg (Phase 2)
Number analyzed (Participants) | 6 | 6 | 14
Participants | 0 | 1 | 3

3. Primary Outcome: Half-life
Description: Mean and standard deviation for the time required for the serum concentration to fall to 50% of its starting dose by dose level and study part.
Time Frame: Prior to, at the end of, and 2 hours after infusion on day 1 of cycles 1-2; days 4 & 8 of cycle 1; prior to and the end of infusion on day 15 of cycle 1; prior to start of infusion on day 15 of cycle 2; prior to start of infusion on day 1 of cycles 3+
Population: all toxicity evaluable patients
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part A: 20 mg/kg (Phase 1) | Part A PK: 20 mg/kg (Expansion) | Part B: 20 mg/kg (Phase 2)
Number analyzed (Participants) | 6 | 6 | 13
hours | 281 (176) | 221 (48) | 162 (64)

4. Primary Outcome: Time to Maximum Concentration (T Max)
Description: Mean and standard deviation for the time at which the maximum (peak) serum concentration occurs by dose level and study part.
Time Frame: as for outcome 3
Population: All toxicity evaluable patients
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part A: 20 mg/kg (Phase 1) | Part A PK: 20 mg/kg (Expansion) | Part B: 20 mg/kg (Phase 2)
Number analyzed (Participants) | 6 | 6 | 13
hours | 1.9 (1.1) | 1.7 (1) | 1.7 (0.9)

5. Primary Outcome: Maximum Concentration (C Max)
Description: Mean and standard deviation for the maximum (peak) serum concentration by dose level and study part.
Time Frame: as for outcome 3
Population: All toxicity evaluable patients
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Part A: 20 mg/kg (Phase 1) | Part A PK: 20 mg/kg (Expansion) | Part B: 20 mg/kg (Phase 2)
Number analyzed (Participants) | 6 | 6 | 13
ug/ml | 175 (78) | 203 (85) | 168 (75)

6. Primary Outcome: Area Under Curve (AUC)
Description: Mean and standard deviation for the area under the drug concentration over time curve by dose level and study part.
Time Frame: as for outcome 3
Population: All toxicity evaluable patients
Measure: Mean (Standard Deviation); unit: hr*ug/ml
Arm/Group | Part A: 20 mg/kg (Phase 1) | Part A PK: 20 mg/kg (Expansion) | Part B: 20 mg/kg (Phase 2)
Number analyzed (Participants) | 6 | 6 | 13
hr*ug/ml | 46913 (29902) | 41328 (9251) | 36811 (17641)

7. Primary Outcome: Clearance
Description: Mean and standard deviation for the rate of elimination of the drug by dose level and study part.
Time Frame: as for outcome 3
Population: All toxicity evaluable patients
Measure: Mean (Standard Deviation); unit: ml/hr
Arm/Group | Part A: 20 mg/kg (Phase 1) | Part A PK: 20 mg/kg (Expansion) | Part B: 20 mg/kg (Phase 2)
Number analyzed (Participants) | 6 | 6 | 13
ml/hr | 40.03 (34.9) | 13.4 (4.6) | 33.2 (25.3)

8. Primary Outcome: Disease Control Rate (Part A)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), no new lesions detected and <20% increase in sum of smallest diameters of lesions; Disease Control Rate = CR + PR + SD
Time Frame: Up to 4 months
Measure: Number; unit: participants
Arm/Group | Part A: 20 mg/kg (Phase 1) | Part A PK: 20 mg/kg (Expansion)
Number analyzed (Participants) | 6 | 6
participants | 0 | 0

9. Primary Outcome: Response (Complete Response or Partial Response) (Part B)
Description: as for outcome 8
Time Frame: Up to 168 days
Measure: Number; unit: participants
Arm/Group | Part B: 20 mg/kg (Phase 2)
Number analyzed (Participants) | 14
participants | 0

10. Secondary Outcome: T-lymphocyte Saturation
Description: Mean and standard deviation for blood samples that will be evaluated for T-lymphocyte saturation by VX15/2503 utilizing a validated flow-cytometry based assay on cycle 1 day 28 (prior to cycle 2 day 1).
Time Frame: Up to 28 days
Population: All Eligible Patients
Measure: Mean (Standard Deviation); unit: percent of T-lymphocyte Saturation
Arm/Group | Part A: 20 mg/kg (Phase 1) | Part A PK: 20 mg/kg (Expansion) | Part B: 20 mg/kg (Phase 2)
Number analyzed (Participants) | 6 | 6 | 14
percent of T-lymphocyte Saturation | 98.06 (3.15) | 99.05 (1.69) | 92.99 (13.79)

11. Secondary Outcome: Total Soluble SEMA4D
Description: Mean and standard deviation of blood and serum samples evaluated for total soluble SEMA4D through a qualified enzyme-linked immunosorbent assay (ELISA) assay.
Time Frame: Up to 28 days
Population: All eligible patients
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Part A: 20 mg/kg (Phase 1) | Part A PK: 20 mg/kg (Expansion) | Part B: 20 mg/kg (Phase 2)
Number analyzed (Participants) | 6 | 6 | 14
pg/mL | 25170.43 (5906.46) | 19757.09 (4680.32) | 25986.81 (7665.71)

12. Secondary Outcome: Immunogenicity of Pepinemab
Description: Mean and standard deviation of immunogenicity assessed in serum through a qualified ELISA.
Time Frame: Up to 3 years
Population: The planned assays for ADA were unable to generate interpretable results due to limitations of the assay which resulted in higher levels of false positive results. These samples were re-run and only one confirmed positive result out of 81 samples, which was considered to be a true positive ADA. Even this one confirmed positive result had a negative titer, which further signifies a possible false positive or very low-level ADA. Therefore, results were determined to be unreliable and invalid.
Arm/Group | Part A: 20 mg/kg (Phase 1) | Part A PK: 20 mg/kg (Expansion) | Part B: 20 mg/kg (Phase 2)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 28 months
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. All-Cause Mortality includes all deaths collected on the study. Ineligible patients are excluded from reporting of adverse events.
Arm/Group | Part A: 20 mg/kg (Phase 1) | Part A PK: 20 mg/kg (Expansion) | Part B: 20 mg/kg (Phase 2)
All-Cause Mortality (participants affected / at risk) | 1/6 | 0/6 | 3/14
Serious Adverse Events (participants affected / at risk) | 4/6 | 4/6 | 10/14
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: 20 mg/kg (Phase 1) (N=6) | Part A PK: 20 mg/kg (Expansion) (N=6) | Part B: 20 mg/kg (Phase 2) (N=14)
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Alkaline phosphatase increased (Investigations) | 0 | 1 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 6
Anorexia (Metabolism and nutrition disorders) | 2 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Creatinine increased (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3
Irregular menstruation (Reproductive system and breast disorders) | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 0 | 5
Mucosal infection (Infections and infestations) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, PROGRESSIVE DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
White blood cell decreased (Investigations) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: 20 mg/kg (Phase 1) (N=6) | Part A PK: 20 mg/kg (Expansion) (N=6) | Part B: 20 mg/kg (Phase 2) (N=14)
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 2
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 2
Agitation (Psychiatric disorders) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 3 | 4
Alkaline phosphatase increased (Investigations) | 6 | 1 | 8
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 5
Anemia (Blood and lymphatic system disorders) | 4 | 4 | 10
Anorexia (Metabolism and nutrition disorders) | 2 | 3 | 7
Anxiety (Psychiatric disorders) | 3 | 1 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 4 | 4
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 8
Blood and lymphatic system disorders - Other, Neutrophil count increased (Blood and lymphatic system disorders) | 0 | 0 | 1
Blood and lymphatic system disorders - Other, RBC decreased (Blood and lymphatic system disorders) | 0 | 0 | 1
Blood and lymphatic system disorders - Other, White Blood Cell Count Increased (Blood and lymphatic system disorders) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Blurred vision (Eye disorders) | 1 | 0 | 1
Body odor (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 2 | 0 | 2
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Chills (General disorders) | 2 | 1 | 4
Cholesterol high (Investigations) | 0 | 1 | 0
Concentration impairment (Nervous system disorders) | 0 | 0 | 1
Confusion (Psychiatric disorders) | 1 | 0 | 2
Constipation (Gastrointestinal disorders) | 2 | 0 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 9
Creatinine increased (Investigations) | 1 | 0 | 1
Cushingoid (Endocrine disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0
Depression (Psychiatric disorders) | 3 | 2 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
Ear and labyrinth disorders - Other, (Ear and labyrinth disorders) | 0 | 0 | 1
Edema limbs (General disorders) | 1 | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1
Eye disorders - Other, Anisocoria (Eye disorders) | 0 | 0 | 1
Eye disorders - Other, Vision decreased (Eye disorders) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fatigue (General disorders) | 3 | 3 | 6
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 1
Fever (General disorders) | 3 | 2 | 10
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 2 | 0
Gait disturbance (General disorders) | 2 | 0 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 2
General disorders and administration site conditions - Other, Generalized edema (General disorders) | 0 | 0 | 1
General disorders and administration site conditions - Other, SWEATING (General disorders) | 1 | 0 | 0
Genital edema (Reproductive system and breast disorders) | 0 | 0 | 1
Gynecomastia (Reproductive system and breast disorders) | 1 | 0 | 0
Hallucinations (Psychiatric disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 3 | 7
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0
Hematuria (Renal and urinary disorders) | 2 | 1 | 2
Hemoglobin increased (Investigations) | 0 | 0 | 2
Hemoglobinuria (Renal and urinary disorders) | 0 | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hot flashes (Vascular disorders) | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 4 | 9
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypertension (Vascular disorders) | 4 | 2 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 1 | 8
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 1 | 5
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1 | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 1 | 2
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 1 | 7
Hypotension (Vascular disorders) | 1 | 2 | 3
Hypothyroidism (Endocrine disorders) | 0 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
INR increased (Investigations) | 0 | 0 | 2
Infusion related reaction (General disorders) | 3 | 2 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 2 | 2
Infusion site extravasation (General disorders) | 1 | 0 | 0
Injury, poisoning and procedural complications - Other, OPEN WOUND (Injury, poisoning and procedural complications) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 0 | 5
Investigations - Other, BICARBONATE LOW (Investigations) | 2 | 0 | 0
Investigations - Other, ELEVATED BICARBONATE SERUM LOW (Investigations) | 1 | 0 | 0
Investigations - Other, ELEVATED LDH (Investigations) | 1 | 0 | 1
Investigations - Other, HYOCHLOREMIA (Investigations) | 0 | 0 | 1
Investigations - Other, HYPOCHLOREMIA (Investigations) | 1 | 0 | 1
Investigations - Other, LDH INCREASED (Investigations) | 1 | 0 | 0
Investigations - Other, LDH increased (Investigations) | 0 | 0 | 1
Investigations - Other, Monocytes Decrease (Investigations) | 0 | 0 | 1
Investigations - Other, Monocytes Increased (Investigations) | 0 | 0 | 1
Investigations - Other, bicarbonate serum low (Investigations) | 0 | 1 | 0
Investigations - Other, elevated BUN (Investigations) | 0 | 1 | 0
Investigations - Other, elevated LDH (Investigations) | 0 | 1 | 0
Irritability (General disorders) | 1 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4
Keratitis (Eye disorders) | 0 | 0 | 1
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 1 | 0
Localized edema (General disorders) | 1 | 0 | 1
Lung infection (Infections and infestations) | 0 | 1 | 1
Lymphocyte count decreased (Investigations) | 0 | 3 | 9
Malaise (General disorders) | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1
Metabolism and nutrition disorders - Other, HYPOCHLOREMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
Metabolism and nutrition disorders - Other, Hyperchloremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Metabolism and nutrition disorders - Other, Increased bicarbonates (Metabolism and nutrition disorders) | 0 | 0 | 1
Metabolism and nutrition disorders - Other, Increased phosphorus level (Metabolism and nutrition disorders) | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal and connective tissue disorder - Other, DIFFICULTY FULLY EXTENDING LEFT LEG (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal and connective tissue disorder - Other, LEFT MEDIAL THIGH SWELLING (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, LIMP (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal and connective tissue disorder - Other, MUSCLE ACHES/PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal and connective tissue disorder - Other, muscle spasm (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 4 | 1 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Nervous system disorders - Other, Spinal cord compression (Nervous system disorders) | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 1 | 3
Non-cardiac chest pain (General disorders) | 1 | 1 | 5
Optic nerve disorder (Eye disorders) | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1
Pain (General disorders) | 2 | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 3 | 6
Paresthesia (Nervous system disorders) | 1 | 1 | 2
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1 | 3
Phantom pain (Nervous system disorders) | 2 | 0 | 0
Photophobia (Eye disorders) | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 6
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Proteinuria (Renal and urinary disorders) | 1 | 2 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Reproductive system and breast disorders - Other, GENITAL HYPERSENSITIVITY (Reproductive system and breast disorders) | 0 | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, HEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, MILD RHINORREA G1 (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, RHINORRHEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 1
Serum amylase increased (Investigations) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 5 | 2 | 7
Skin and subcutaneous tissue disorders - Other, FACIAL SORES (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, FISTULA - SUPERIOR LATERAL STUMP WOUND (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, MOTTLING OF FINGERS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, SEBORRHEIC DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, Skin breakdown (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 2 | 1 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 2
Upper respiratory infection (Infections and infestations) | 0 | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 2
Urinary urgency (Renal and urinary disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 1 | 4
Weight gain (Investigations) | 0 | 1 | 1
Weight loss (Investigations) | 2 | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
White blood cell decreased (Investigations) | 2 | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior sponsor approval

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/30/NCT03320330/Prot_SAP_000.pdf